CLINICAL TRIAL: NCT03433027
Title: A Phase 2 Trial of Intratumoral EGFR Antisense DNA (BB-401) in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (HNSCC) Who Have Failed All Available Standard Therapies
Brief Title: A Study of BB-401 in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benitec Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BB-401-01
Record Dates: First submitted 2018-02-05; First posted 2018-02-14 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BB-401 (Experimental): BB-401 Intratumoral injection
  Interventions: Drug: BB-401

INTERVENTIONS:
Drug: BB-401 — BB-401 1.92ug/mL Intratumoral Injections, every week for up to 8 weeks

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of intratumoral injections with an Epidermal Growth Factor Receptor (EGFR) AntiSense DNA (BB-401) in patients with metastatic/recurrent HNSCC.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed HNSCC
* Failed (or are ineligible/decline to receive) all available standard therapies
* Stable, treated brain metastases
* One target lesion defined as measurable (via RECIST v1.1), with a maximum longest diameter of 4 cm, and suitable for injection
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Agree to biopsies of a selected primary lesion and where possible of a second untreated lesion at baseline and end of treatment
* Ceased anti-cancer therapy for at least 3 weeks or 5 half-lives for chemotherapy based treatment regimen, or 4 weeks from any therapy with therapeutic biologicals or any type of investigational therapy

Key Exclusion Criteria:

* Nasopharyngeal Carcinoma
* Concomitant anti-cancer therapy
* Unresolved toxicities from prior treatments
* Patients in whom the indicator lesion is at risk of hemorrhage or clinically significant swelling/inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
Overall Response (OR) of the injected tumor | Up to 20 months (estimated length of the study)
  Overall response is defined as Complete Response (CR) or Partial Response (PR) as evaluated using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee version 1.1

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | End of Treatment Visit (Week 9) through to study end (up to 18 months)
  DCR is measured on a subset of subjects who achieve Stable Disease (SD), Partial Response (PR) or Complete Response (CR) at the End of Treatment visit. DCR will be defined as the proportion of these subjects that show absence of disease progression as evaluated using the RECIST v1.1 criteria
Progression Free Survival (PFS) | Up to 20 months (estimated length of study)
  PFS will be defined as the time from first treatment administration to first observation of documented disease progression as evaluated using the RECIST v1.1 criteria
Overall Survival (OS) | Up to 20 months (estimated length of study)
  OS will be defined as the time from first treatment administration through to death due to any cause
Duration of Response (DoR) | 20 months (estimated length of study)
  DoR assessments will be performed on the subset of patients for who a CR, PR, or SD response is achieved. DoR will be measured from the time where the response criteria are first met, until the first date that progressive disease is objectively documented, or the date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (2):
  - The Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Calvary Central Districts Hospital, Elizabeth Vale, South Australia
- Russia (4):
  - Irkutsk Oncology Center, Irkutsk
  - Clinical Oncology Dispensary #1, Krasnodar
  - Leningrad Regional Oncology Dispensary, Leningrad Region
  - Saint Petersburg City Oncology Clinic, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for primary and secondary outcome measures will be made available for the Interim Analysis and routinely through-out the study for the Data Safety Monitoring Board
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be available within 6-8 weeks from data cut off/lock
Access Criteria: Data will only be available to the Data Safety Monitoring Board and Interim Analysis members